CLINICAL TRIAL: NCT06867367
Title: REducing pSychological diSTress To Optimize Recovery of Elderly ICU Survivors and Caregivers (RESTORE-ICU): A Pilot Feasibility Study
Brief Title: REducing pSychological diSTress To Optimize Recovery of Elderly ICU Survivors and Caregivers (RESTORE-ICU)
Acronym: RESTORE-ICU
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Beth Israel Deaconess Medical Center (Other)
Responsible Party: Principal Investigator, Somnath Bose, MD, Assistant Professor of Anesthesia, Beth Israel Deaconess Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 2024P000984
Record Dates: First submitted 2025-02-26; First posted 2025-03-10 (Actual); Last update posted 2025-06-05 (Actual); Status verified 2025-03

CONDITIONS: Relationship, Family; Well-Being, Psychological
Keywords: mental health; relationship quality; ICU recovery
MeSH Terms: conditions — Psychological Well-Being

STUDY DESIGN:
Intervention Model Description: This is a single-group interventional study in which ICU survivor-caregiver dyads participate in Inner Engineering (IE) practices, including guided meditation (Isha Kriya) and a breathing technique (Nadi Shuddhi). All participants receive the same intervention, delivered via a mobile app or group sessions. The study assesses psychological well-being, relationship quality, and neurological effects using EEG recordings
Masking Description: There is no masking in this study. All participants (caregiver-patient dyads) are aware of the intervention they are receiving (Inner Engineering practices, including Isha Kriya and Nadi Shuddhi)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Arm 1 (Experimental): This arm involves ICU survivor-caregiver dyads engaging in the Inner Engineering (IE) intervention, including Isha Kriya (15-minute guided meditation) and Nadi Shuddhi (3-5 minute alternate-nostril breathing). The intervention is delivered through a mobile app or group sessions. Participants will complete surveys and EEG recordings to assess changes in psychological well-being, relationship quality, and neural activity. Both patients and caregivers will be introduced to the interventions either remotely or in-person, followed by remote delivery via the 3Cs app. The app tracks usage metrics.
  Nadi Shuddhi - A 4-minute breathing practice for mental balance and relaxation, to be practiced daily.
  Isha Kriya - A 15-minute meditation incorporating breath and awareness, to be practiced at least once (ideally twice) daily
  Interventions: Behavioral: Isha Kriya and Naddi Shuddhi

INTERVENTIONS:
Behavioral: Isha Kriya and Naddi Shuddhi — Isha Kriya, a 15-minute guided meditation, and Nadi Shuddhi, a 3-5-minute alternate-nostril breathing practice. Participants in the intervention groups will be instructed to practice ideally twice or at least once daily.

SUMMARY:
This research study aims to explore whether a set of simple breathing techniques and guided meditations can improve the psychological well-being and recovery of ICU survivors and their caregivers.

ICU survivors and their caregivers often experience high levels of stress, anxiety, and depression after discharge. This study investigates whether practicing Isha Kriya, a guided meditation, and Nadi Shuddhi, a breathing technique, can support their mental health and relationship quality. These practices are delivered through a mobile app or in a group setting.

Participants enroll as a caregiver-patient dyad and will engage in these techniques throughout the study. In addition to the practices, brain activity will be recorded using a safe, non-invasive EEG device. The EEG, a lightweight cap with small sensors, measures brainwaves to assess potential changes in brain function and connection. EEG recordings will take place in the hospital during two sessions, each lasting approximately 40 minutes.

Participants will also complete short surveys at five time points throughout the study, assessing mood, stress, and relationship quality. Baseline demographic information will be collected, and at the conclusion of the study, a brief interview will be conducted to gather feedback on the experience.

The study spans approximately seven weeks, with the overall goal of determining whether these breathing and meditation practices can provide accessible and scalable mental health support for ICU survivors and their caregivers.

DETAILED DESCRIPTION:
Overview of the Study This study will evaluate the feasibility of implementing a mindfulness-based intervention, Inner Engineering (IE) practices, with concurrent EEG measurements among elderly ICU survivors aged 60 to 85 years and their caregivers. The intervention includes Isha Kriya and Nadi Shuddhi, two simple and accessible meditation practices delivered via a secure digital platform. The study aims to assess feasibility, acceptability, and barriers to implementation while testing paired EEG hyperscanning to explore neural congruency between participants. Conducted in two phases, the study will refine the research infrastructure and optimize the delivery of IE practices, first in the hospital setting and then remotely in home environments.

Overall Study Design This proof-of-concept pilot study utilizes an interventional, mixed-methods design combining experimental feasibility testing, EEG hyperscanning, and qualitative assessments. The study is divided into two phases: Phase 1 focuses on refining infrastructure for delivering IE and EEG monitoring in the hospital, while Phase 2 transitions to evaluating the feasibility of remote intervention delivery and monitoring in participants' homes.

Intervention Isha Kriya, a 15-minute guided meditation, and Nadi Shuddhi, a 3-5-minute alternate-nostril breathing practice. Participants in the intervention groups will be instructed to practice ideally twice or at least once daily. The study interventions will be introduced in-person for patients and either in-person or remotely for their caregivers. After the initial introduction, the interventions will be administered via the 3Cs app. This application has been used for meditation interventions and allows accurate tracking of usage metrics.

Nadi Shuddhi - a gentle 4-minute breathing practice for creating mental balance and relaxation, to be practiced for a minimum of 4 minutes daily.

https://www.youtube.com/watch?v=q5m6tMjcF8k

Isha Kriya - a 15-minute guided meditation that incorporates the breath and the awareness to create mental clarity and health, to be practiced at least once (ideally twice) daily. https://www.youtube.com/watch?v=EwQkfoKxRvo

Phase 1: Refining Hospital-Based Procedures Phase 1 focuses on establishing the research infrastructure within the hospital setting to optimize the implementation of Inner Engineering (IE) practices and EEG hyperscanning. Two ICU survivor-caregiver dyads will be recruited, with survivors defined as individuals aged 60-85 years who experienced an ICU stay of five or more days, and caregivers who self-identify as such and either live with or frequently visit the survivor. Baseline data collection will include high-fidelity EEG hyperscanning and psychological surveys. After learning and practicing IE, participants will complete another EEG hyperscanning data collection and post-intervention assessments. Semi-structured interviews will provide critical feedback on the intervention's acceptability and feasibility, helping to refine study processes for future phases.

Phase 2: Post-Discharge Implementation Phase 2 evaluates the feasibility of implementing IE practices after hospital discharge, focusing on participants' adherence to daily meditation practices. Five ICU survivor-caregiver dyads will be enrolled. At the hospital, baseline data collection will include EEG hyperscanning with the high-density R-Net system and psychological surveys. Participants will then learn the IE practices, with instructions to practice ideally twice or at least once daily. Post-intervention data will be collected afterwards, including EEG hyperscanning and surveys. After discharge to home, participants will be instructed to practice surveys will be completed at weeks 2, 4, and 6. At the end of week 6, a semi-structured interview will gather feedback on the intervention's feasibility, acceptability, and barriers to enrollment or retention.

ELIGIBILITY:
Patient Inclusion/Exclusion Criteria

Inclusion Criteria:

1. Provide signed and dated informed consent and understand the nature of the study sufficiently to allow completion of all study assessments.
2. Elderly ICU survivors aged over 60 years who have experienced long ICU stays of more than five days.
3. Caregivers who either live in the same household as the survivor or visit more than three times a week.

Exclusion Criteria:

Co-enrollment in other interventional studies will not be allowed.

1. Age >=85 years (Justification: Assessment instruments not validated in this age group and patients in extremes of age may have limited proficiency to engage in proposed meditative practices)
2. Non-English speaking/Low-English proficiency (Justification: assessment instruments are not validated in a sufficient range of languages, and the research team lacks polylingual capabilities or the financial resources to hire interpreters for the duration of all proposed assessments.)
3. Non-US resident
4. Recent or current meditation, yoga, breathwork or associated MBI intervention practice (> 2 times per week). (Justification: as the primary outcome is to evaluate the feasibility and adherence of patients to a multicomponent MBI, recent or current practice of the individual or combined components would directly influence the endpoint).
5. Individuals discharged to a non-home location, such as a rehabilitation center, nursing home, or long-term acute care facility.
6. Individuals with limited internet access, which would prevent access to online guided meditation
7. Prisoners.
8. Individuals who refuse to participate in the study.
9. Not on vasopressor or inotropic support at the time of enrollment.
10. Not on non-invasive ventilation, high-flow nasal cannula (HFNC), or mechanically ventilated.
11. Not on continuous renal replacement therapy (CRRT).
12. Failure to pass Informant Questionnaire on Cognitive Decline in the Elderly (IQCODE) screening (>3.6; Justification: Cognitive decline would limit the ability to engage with and complete the study interventions and assessments).
13. Scores ≥ 5 on either the anxiety or depression subscales suggesting severe symptom levels.
14. Known diagnosis of moderate or severe dementia.
15. Neurological injury.
16. Residing in a medical institution before admission.
17. Patient on hospice at or before the time of enrollment.
18. Mechanical ventilation at baseline or solely for airway protection.
19. Patient not expected to go home (e.g., transfer to a facility).
20. Patient not expected to survive two months or expected to transition to hospice.
21. Patient died in hospital before enrollment.
22. Attending physician declined enrollment.
23. Patient discharged before being approached for consent.
24. Either the patient or caregiver in the dyad declined participation (based on IQCODE or consent).

Caregiver Inclusion/Exclusion Criteria

Inclusion Criteria:

1. Provide signed and dated informed consent and understand the nature of the study sufficiently to allow completion of all study assessments.
2. Caregivers who either live in the same household as the survivor or visit more than three times a week.
3. Age ≥18 years old.

Exclusion Criteria:

1. Non-English speaking/Low-English proficiency (Justification: assessment instruments are not validated in a sufficient range of languages, and the research team lacks polylingual capabilities or the financial resources to hire interpreters for the duration of all proposed assessments.)
2. Non-US resident
3. Recent or current meditation, yoga, breathwork or associated MBI intervention practice (> 2 times per week). (Justification: as the primary outcome is to evaluate the feasibility and adherence of patients to a multicomponent MBI, recent or current practice of the individual or combined components would directly influence the endpoint).
4. Individuals with limited internet access, which would prevent access to online guided meditation
5. Prisoners.
6. Individuals who refuse to participate in the study.
7. Diagnosed with severe psychiatric disorders, such as schizophrenia, bipolar disorder, or ongoing substance abuse, that could interfere with participation.
8. Individuals actively receiving treatment for recent trauma
9. Scores ≥ 5 on either the anxiety or depression subscales suggesting severe symptom levels.
10. severe or acute medical illness

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 14 (Estimated)
Dates: Start 2025-07 (Estimated); Primary Completion 2025-08 (Estimated); Study Completion 2025-10 (Estimated)

PRIMARY OUTCOMES:
Participant Adherence to the Inner Engineering (IE) Intervention | 7 weeks (from baseline assessment to post-intervention follow-up)
  Adherence will be assessed based on the number of IE sessions each participant completes.
Participant Engagement with the Inner Engineering (IE) Intervention | 7 weeks (from baseline assessment to post-intervention follow-up)
  Engagement will be measured by the frequency of practice logged in the mobile app, indicating participant involvement in the intervention.
Study Retention Rate | 7 weeks (from baseline assessment to post-intervention follow-up)
  Retention will be assessed by tracking the percentage of participants who complete the full study period, including all study assessments.

SECONDARY OUTCOMES:
Changes in Perceived Stress | 7 weeks (baseline, weeks 2, 4, and 6 post-intervention)
  Changes in perceived stress will be assessed using the Perceived Stress Scale (PSS) to measure perceived stress levels. The PSS ranges from 0 to 40, with higher scores indicating higher levels of perceived stress.
Changes in Psychological distress related to traumatic events | 7 weeks (baseline, weeks 2, 4, and 6 post-intervention)
  Changes in Psychological distress related to traumatic events will be assessed using the Impact of Event Scale-Revised (IES-R). The IES-R ranges from 0 to 88, with higher scores indicating greater levels of distress related to traumatic events.
Changes in Anxiety and Depressive symptoms | 7 weeks (baseline, weeks 2, 4, and 6 post-intervention)
  Changes in anxiety and depressive symptoms will be assessed using the Patient Health Questionnaire-4 (PHQ-4). The PHQ-4 ranges from 0 to 12, with higher scores indicating higher levels of depressive symptoms and anxiety.
Changes in Caregivers' Interpersonal Connection | 7 weeks (baseline, weeks 2, 4, and 6 post-intervention)
  Caregivers' Interpersonal connection will be assessed using the Interpersonal Mindfulness Scale (IMS). The IMS total score involves reverse scoring indicated items and calculating the mean score (between 1 to 5). Higher scores indicate greater mindfulness and interpersonal connection.
Changes in Caregivers' Compassion for Self and Others | 7 weeks (baseline, weeks 2, 4, and 6 post-intervention)
  Caregiver's compassion for self and others will be assessed using the Compassion for Self and Others Scale (CS). The total score involves reverse scoring indicated items and calculating the mean score (between 1 to 5). Higher scores indicate greater compassion for self and others.
Changes in Relationship Quality | 7 weeks (baseline, weeks 2, 4, and 6 post-intervention)
  Relationship quality between caregivers and patients between patients and caregivers will be assessed using the Dyadic Relationship Scale (DRS). The DRS includes two subscales: dyadic strain and positive dyadic interaction, which are measured using a four-option response scale (1 to 4). Higher scores on both subscales indicate higher levels of dyadic strain or positive dyadic interaction, respectively.

CONTACTS AND LOCATIONS:
Locations (1):
- Beth Israel Deaconess Medical Center, Boston, Massachusetts, United States